CLINICAL TRIAL: NCT03719248
Title: High Thoracic Epidural Reduces Risks of Increased Left Ventricular Mass Index and Coronary Vascular Disease During Aortic Valve Replacement Alone or in Addition to Coronary Artery Bypass Graft Surgery
Brief Title: Thoracic Epidural Reduces Risks of Increased Left Ventricular Mass Index During Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Said Elgebaly,MD (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Said Elgebaly,MD, director, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TantaU
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Ischemia Coronary Artery Origin
Keywords: Epidural.; ventricular mass; Aortic valve; coronary bypass
MeSH Terms: interventions — Echocardiography; Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- HTEA Group + N(LVMI)+ AVR alone(n=10) (Active Comparator): HTEA Group + N(LVMI)+ AVR alone(n=10)
  Interventions: Device: thoracic epidural
- HTEA Group + ↑ (LVMI)+ AVR alone(n=10) (Active Comparator): HTEA Group + ↑ (LVMI)+ AVR alone(n=10)
  Interventions: Device: thoracic epidural
- HTEA Group + N(LVMI)+ AVR + CABG(n=10) (Active Comparator): HTEA Group + N(LVMI)+ AVR + CABG(n=10)
  Interventions: Device: thoracic epidural
- HTEA Group +↑ (LVMI)+ AVR + CABG(n=10) (Active Comparator): HTEA Group +↑ (LVMI)+ AVR + CABG(n=10)
  Interventions: Device: thoracic epidural
- Control(GA) Group+ N(LVMI)+ AVR alone(n=10) (No Intervention): Control(GA) Group+ N(LVMI)+ AVR alone(n=10)
- Control(GA) Group+ ↑ (LVMI)+ AVR alone(n=10) (No Intervention): Control(GA) Group+ ↑ (LVMI)+ AVR alone(n=10)
- Control(GA) Group+ N(LVMI)+ AVR + CABG(n=10) (No Intervention): (GA) Group+ N(LVMI)+ AVR + CABG(n=10)
- Control(GA) Group+↑ (LVMI)+ AVR + CABG(n=10) (No Intervention): Control(GA) Group+↑ (LVMI)+ AVR + CABG(n=10)

INTERVENTIONS:
Device: thoracic epidural — high thoracic epidural anesthesia (HTEA) combined with GA, transesophageal, transthoracic echocardiography and Holter ECG
  Other Names: high thoracic epidural anesthesia (HTEA) combined with GA; transesophageal and transthoracic echocardiography; Holter ECG
  Arms: HTEA Group + N(LVMI)+ AVR + CABG(n=10); HTEA Group + N(LVMI)+ AVR alone(n=10); HTEA Group + ↑ (LVMI)+ AVR alone(n=10); HTEA Group +↑ (LVMI)+ AVR + CABG(n=10)

SUMMARY:
Increased left ventricular mass index (LVMI) results from aortic valve lesions as an adaptive mechanism to help limit systolic wall stress and preserve ejection fraction (EF). This study Aim to investigate the effects of sympathetic blockade by HTEA on systolic and diastolic LV function in patients undergoing aortic valve replacement (AVR) alone or in addition to coronary artery bypass graft (CABG). It Designs as A prospective randomized controlled comparative study in which eighty patients received either general anesthesia ( control group n=40) or with high thoracic epidural analgesia(HTEA group n=40). Each group subdivided to normal (LVM) (n=20)or increased(LVM) group(n=20), all submitted to (AVR) alone or in addition to (CABG).

DETAILED DESCRIPTION:
Background: Increased left ventricular mass index (LVMI) results from aortic valve lesions as an adaptive mechanism to help limit systolic wall stress and preserve ejection fraction (EF).

Aim: to investigate the effects of sympathetic blockade by HTEA on systolic and diastolic LV function in patients undergoing aortic valve replacement (AVR) alone or in addition to coronary artery bypass graft (CABG).

Design: A prospective randomized controlled comparative study. Methods: Eighty patients received either general anesthesia ( control group n=40) or with high thoracic epidural analgesia(HTEA group n=40). Each group subdivided to normal (LVM) (n=20)or increased(LVM) group(n=20), all submitted to (AVR) alone or in addition to (CABG).Perioperative heart rate (HR), mean arterial blood pressure (MAP), incidence of ischemic ECG, LV systolic and diastolic function changes were measured till 48 h, postoperatively.

Patients were subjected to ambulatory Holter monitoring, Hemodynamic measures, intraoperative transesophageal echocardiography (iTEE) and postoperative Trans Thoracic Echocardiography (TTE) to assess myocardial ischemia and Left ventricular systolic/diastolic function.

ELIGIBILITY:
Inclusion Criteria:

* patients between 65 and 75 years with:
* physical status of ASA II and IV
* who underwent aortic valve replacement (for isolated or mixed aortic valve lesions) alone or in addition to-coronary artery bypass grafting. in the Cardio-thoracic Surgery Department of Tanta University Hospital during a two year period were enrolled in this study.
* Before inclusion in the study, all patients were evaluated with extended echocardiographic imaging, full history including cardiac symptoms (dyspnea, orthopnea, paroxysmal nocturnal dyspnea, chest pain, and low cardiac output symptoms) was taken from all patients. General (including body weight and height) and systematic (including cardiac examination) examinations were done to all patients.

Exclusion Criteria:

* Patients with an ejection fraction of 0.3, myocardial infarction within the last 4 weeks
* diabetes
* severe pulmonary or arterial hypertension.
* a contraindication for HTEA.
* patients without preoperative optimal echocardiographic imaging were excluded.
* Among the exclusion criteria were the administration of ticlopidine within 15 days before surgery and the administration of platelet glycoprotein IIb/IIIa inhibitors. In common with previous investigators, we did not consider treatment with low-molecular-weight heparin and aspirin below the dosage of 160 mg/day to be contraindications to the procedure.
* Patients with significant aortic insufficiency were also excluded from the study in order to avoid introducing further variables that could influence hemodynamic response to the procedure.
* Patients were excluded if they underwent an AVR on an emergency basis, had poor acoustic windows for adequate echocardiographic assessment, and/or did not undergo an echocardiogram before the operation.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
The changes in LV systolic. | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively.
  LV end systolic diameter (LVESD)
The changes in LV diastolic. | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively.
  Left ventricular end diastolic diameter (LVEDD)
ejection fraction percent | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively.
  changes in percentage, of how much blood the left ventricle pumps out with each contraction.
FAC percent | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively.
  Fractional Area Change (FAC) percent
  Fractional Area Change (FAC)
EDA | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively.
  end-diastolic area (EDA)

SECONDARY OUTCOMES:
Perioperative changes in heart rate (HR). | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively
  during evaluation of hemodynamic changes.
changes in mean arterial blood pressure (MAP) | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively
  during evaluation of hemodynamic changes.
the changes incidence of ischemic ECG. | 5 minutes pre-operatively, 5 minutes after induction of anesthesia,15 minutes before,15 minutes after bypass and at 6, 12, 24 and 48 hour, postoperatively
  Holter monitor tapes were analyzed for myocardial ischemia based the criteria of horizontal or down-sloping ST-segment depression of > 1 mm below the baseline, lasting for at least 1 min. Events were separated by at least 5 min without ECG ischemia ECG changes included new ST-T changes, T inversion, Q waves and/or a bundle branch block

CONTACTS AND LOCATIONS:
Overall Officials: ahmed S Elgebaly, MD, Principal Investigator — assist .professor
Locations (1):
- Ahmed Said Elgebaly, Tanta, Egypt

REFERENCES:
- [Result] Schmidt C, Hinder F, Van Aken H, Theilmeier G, Bruch C, Wirtz SP, Burkle H, Guhs T, Rothenburger M, Berendes E. The effect of high thoracic epidural anesthesia on systolic and diastolic left ventricular function in patients with coronary artery disease. Anesth Analg. 2005 Jun;100(6):1561-1569. doi: 10.1213/01.ANE.0000154963.29271.36. PMID 15920175
- [Result] Berendes E, Schmidt C, Van Aken H, Hartlage MG, Wirtz S, Reinecke H, Rothenburger M, Scheld HH, Schluter B, Brodner G, Walter M. Reversible cardiac sympathectomy by high thoracic epidural anesthesia improves regional left ventricular function in patients undergoing coronary artery bypass grafting: a randomized trial. Arch Surg. 2003 Dec;138(12):1283-90; discussion 1291. doi: 10.1001/archsurg.138.12.1283. PMID 14662525
- [Result] Blomberg S, Emanuelsson H, Kvist H, Lamm C, Ponten J, Waagstein F, Ricksten SE. Effects of thoracic epidural anesthesia on coronary arteries and arterioles in patients with coronary artery disease. Anesthesiology. 1990 Nov;73(5):840-7. doi: 10.1097/00000542-199011000-00008. PMID 2240673
- [Result] Svircevic V, Nierich AP, Moons KG, Diephuis JC, Ennema JJ, Brandon Bravo Bruinsma GJ, Kalkman CJ, van Dijk D. Thoracic epidural anesthesia for cardiac surgery: a randomized trial. Anesthesiology. 2011 Feb;114(2):262-70. doi: 10.1097/ALN.0b013e318201d2de. PMID 21239976
- [Result] Conrady AO, Rudomanov OG, Zaharov DV, Krutikov AN, Vahrameeva NV, Yakovleva OI, Alexeeva NP, Shlyakhto EV. Prevalence and determinants of left ventricular hypertrophy and remodelling patterns in hypertensive patients: the St. Petersburg study. Blood Press. 2004;13(2):101-9. doi: 10.1080/08037050410031855. PMID 15182113
- [Result] Guarracino F, Cariello C, Tritapepe L, Doroni L, Baldassarri R, Danella A, Stefani M. Transoesophageal echocardiography during coronary artery bypass procedures: impact on surgical planning. HSR Proc Intensive Care Cardiovasc Anesth. 2010;2(1):43-9. PMID 23440403
- [Result] El-Morsy GZ, El-Deeb A. The outcome of thoracic epidural anesthesia in elderly patients undergoing coronary artery bypass graft surgery. Saudi J Anaesth. 2012 Jan;6(1):16-21. doi: 10.4103/1658-354X.93048. PMID 22412771
- [Result] Crescenzi G, Landoni G, Monaco F, Bignami E, De Luca M, Frau G, Rosica C, Zangrillo A. Epidural anesthesia in elderly patients undergoing coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2009 Dec;23(6):807-12. doi: 10.1053/j.jvca.2009.02.003. Epub 2009 Apr 19. PMID 19376734
- [Result] Devereux RB, Reichek N. Echocardiographic determination of left ventricular mass in man. Anatomic validation of the method. Circulation. 1977 Apr;55(4):613-8. doi: 10.1161/01.cir.55.4.613. PMID 138494
- [Result] Orsinelli DA, Aurigemma GP, Battista S, Krendel S, Gaasch WH. Left ventricular hypertrophy and mortality after aortic valve replacement for aortic stenosis. A high risk subgroup identified by preoperative relative wall thickness. J Am Coll Cardiol. 1993 Nov 15;22(6):1679-83. doi: 10.1016/0735-1097(93)90595-r. PMID 8227838